CLINICAL TRIAL: NCT05675358
Title: Virtual Reality on Pain, Fear, and Emotional Appearance During Phlebotomy in Pediatric Hematology and Oncology Patients
Acronym: VR-PHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, pHD, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ASBU 2022/89
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Virtual Reality; Pain, Acute; Pediatric Cancer
Keywords: virtual reality; phlebotomy; pain; fear; anxiety; emotional apperance
MeSH Terms: conditions — Acute Pain; Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The child's pain and fear were evaluated blindly to each other by the parent and the nurse who performed the phelobotomy attempt.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): In the study, Oculus Quest 2 256 GB All-In-One Vr Virtual Reality Glasses were used, and the Epic Roller Coasters train game, an application that would attract the attention of children, was determined by the researchers. The virtual reality application was started 2 minutes before the procedure and continued until the procedure was completed.
  Interventions: Behavioral: Virtual Reality
- control (No Intervention): The child in the control group did not receive any additional intervention.

INTERVENTIONS:
Behavioral: Virtual Reality — Oculus Quest 2 256 GB All-In-One Vr Virtual Reality Glasses were used in the study.
  Arms: virtual reality

SUMMARY:
In this study, the effect of virtual reality, which is one of the pain relief methods, on the pain, fear and emotional appearance associated with the procedure, was evaluated in children aged 4-12 years who will undergo phelobotomy in a Pediatric Hematology and Oncology outpatient clinic.

DETAILED DESCRIPTION:
This prospective randomized controlled study was conducted in the pediatric hematology and oncology polyclinic blood collection unit of a university hospital in Turkey.

Patients undergoing phelobotomy were allocated to virtual reality or control groups according to a stratified randomization scheme.

ELIGIBILITY:
Inclusion Criteria:

the age range is between 4-12

to apply to the pediatric hematology and oncology outpatient clinic and to have blood taken

consent of the child and parent to voluntarily participate in the study

The child does not have a physical or psychological deficit that would prevent them from wearing glasses to watch virtual reality.

Exclusion Criteria:

having a fever (>37.5C) and severe dehydration

Before the invasive procedure, the patient was given anagesics.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | procedure - during the phelobotomy
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10
Fear assesed by Child Fear Scale | procedure -during the phelobotomy
  The Child Fear Scale (CFS), this one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear.
Anxiety assesed by Children Anxiety Meter-State | procedure- during the phelobotomy
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10).

SECONDARY OUTCOMES:
emotional apperance assesed by Emotional Appearance Scale for Children | Baseline - before the phelobotomy
  This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'.
  Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, pHD, RN, Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Kanad N, Ozalp Gerceker G, Eker I, Sen Susam H. The effect of virtual reality on pain, fear and emotional appearance during blood draw in pediatric patients at the hematology-oncology outpatient clinic: A randomized controlled study. Eur J Oncol Nurs. 2024 Feb;68:102495. doi: 10.1016/j.ejon.2023.102495. Epub 2023 Dec 26. PMID 38184927